CLINICAL TRIAL: NCT07057453
Title: National Childhood Obesity Prevention Programme BE FIT 24
Acronym: BE FIT 24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Czech Technical University in Prague (Other); STOB CZ s.r.o. (Unknown); Charles University, Czech Republic (Other); Ceska Lekarska Spolecnost Jana Evangelisty Purkyne z.s. (Other); Czech Medical Chamber (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UZIS 2025/5
Record Dates: First submitted 2025-05-23; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Childhood Obesity
Keywords: Early detection; Overweight; Fitness bracelets
MeSH Terms: conditions — Pediatric Obesity; Overweight | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Overweight Children (Other): Overweight children aged 6-11 years who will receive a fitness bracelet and use a gamified mobile app to encourage physical activity and healthy habits through interactive challenges and rewards.
  Interventions: Other: Motivation Engagement for Movement and Interactive Nutrition Development

INTERVENTIONS:
Other: Motivation Engagement for Movement and Interactive Nutrition Development — The intervention includes using of fitness bracelets, a gamified mobile app, a web portal, and regular pediatric check-ups to support healthy habits in overweight children (6-11 years). The bracelets track physical activity, while the mobile app monitors energy balance, encouraging movement and healthy eating through challenges and rewards. The web portal provides family education, and pediatric check-ups track progress and overall health outcomes.

SUMMARY:
The project is a national, prospective, multicenter, interventional pilot project of early detection of childhood overweight and the prevention of obesity in the Czech Republic.

The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure of early detection of childhood overweight and the prevention of obesity and setting up and testing new methods and implementation into the system of health care.

DETAILED DESCRIPTION:
The project is a national, prospective, multicenter, interventional pilot project of early detection of childhood overweight and the prevention of obesity in the Czech Republic.

The aim of the project is to prepare and test innovative tools for optimization of health parameters in childhood, including the preparation of a general health prevention program for obesity as one of the main predeterminants of negative health development in the child population. The primary measurable clinical goal of the project is a 5% reduction in Body mass index (BMI) in children after completing the one-year program.

The project will engage approximately 1,000 overweight children aged 6-11 years in an innovative, gamified experience promoting a healthy lifestyle. Each child will receive a fitness bracelet to monitor their physical activity, while a fun, interactive mobile app will motivate them through challenges and games to maintain a balanced energy level. Additionally, the whole family will benefit from educational resources on a web portal, encouraging a playful and supportive approach to adopting healthier habits together.

The project is supported by the European Social Fund (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0003842.

Study is conducted at approximately 100 sites across Czechia. For a complete list of study sites, please contact the overall study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-11 years
* BMI: Between the 90th and 97th percentile
* Signed consent to participate in the project and GDPR

Exclusion Criteria:

* Children with a BMI between the 90th and 97th percentile with an associated chronic disease requiring continuous pharmacological treatment

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change in BMI of children over the intervention period | Up to 1 year from enrollment

SECONDARY OUTCOMES:
Changes in BMI by subgroups of children (by gender, age, region, with/without playmate) | Up to 1 year from enrollment
Evaluation of energy expenditure (kilojoules) measured using a fitness bracelet during the competition weeks. | Up to 1 year from enrollment
Proportion of children who completed the full process (one-year participation in the program) | Up to 1 year from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Petr Jehlička, PhD, Study Director — Pediatric Cardiology, Plzeň, Czech Republic
Locations (1):
- Czech Medical Chamber, Prague, Czechia, Czechia